CLINICAL TRIAL: NCT05904431
Title: The Effect of Cognitive Performance on Physical Performance in Adolescent Basketball Players
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, NAİME ULUG, PhD, Atılım University
Other Study IDs: E-59394181-604.01.02-32301
Record Dates: First submitted 2023-05-24; First posted 2023-06-15 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cognitive Performance; Physical Performance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine the relationship between physical fitness parameters and cognitive performance levels in basketball players. It has been shown in the literature that exercise has an effect on cognitive factors. However, there is a limited number of studies examining the relationship between physical performance parameters and cognitive performance in basketball players.

DETAILED DESCRIPTION:
Forty-nine male basketball players aged 14-18 years were included in the study. Vertical jump, agility t, reactive agility, 20 m sprint and Y-shaped balance test were applied to all cases as physical performance tests. Right/left discrimination (Recognise application), two-point discrimination, Stroop Test were applied as cognitive performance tests, and the level of pain threshold was evaluated. In the reactive agility test, reactive response speed was evaluated by using visual stimuli, camera and photocell doors. Pearson correlation analysis was used as statistical analysis method.

ELIGIBILITY:
Inclusion Criteria:

* Male basketball players between the ages of 14-18,
* To be a licensed athlete for at least 5 years,
* Being active in sports and training for the last 1 year,
* Weekly training intensity is at least 5 hours per week

Exclusion Criteria:

* Having a history of visual, mental or systemic disease,
* Having a history of major injury in the medical history,
* Any complaints of acute or chronic pain/injury

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Professional Basketball Athletes
Sampling Method: Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Reactive Agility | 25 June 2023
  For the test, the athletes were positioned in the middle of the distance of 16 feet (4.88 meters), 2 meters in front of the warning screen. A and B funnels were introduced to the athlete. When the test started, the warning screen started counting down from 3; at the end of the count, it gave one of the warnings A or B as a random warning. As soon as the athlete saw the warning, he started the test in the direction of the warning that appeared on the screen. The time elapsed between the appearance of the A or B warning on the screen and the athlete's perception and response (knee flexion) was recorded as "reaction time" by watching the Movavi Video Editor Plus 2022 program. After starting the test, the athlete ran and touched the first funnel he turned to, then came back and touched the other funnel. . He turned back to the funnel he touched first and passed through the photocells, completing the test. The time from start to finish was recorded as "reactive agility score".
Lower Extremity Strength | 25 June 2023
  Microgate Witty Brand vertical jump mat was used to evaluate the vertical jump height. The device consists of 2 parts, a matte and a tablet. For the test, the athlete was asked to jump on the mat as described. When the athlete performed the vertical jump, the jump height was recorded by reading from the tablet screen. Before the test, the athletes were given 2 repetitive vertical jumps for trial purposes.
Agility | 25 June 2023
  Agility T Test was used to evaluate Agility. The T-Test was performed using a standardized version from the previous literature [65]. A 10 × 10 meter course was created for the test. The funnels defining the boundaries of the track were numbered. Athletes were asked to return to the cone alignments according to the order specified for the test.
Running Speed | 25 June 2023
  The 20-meter sprint test was used to evaluate the running speed. A 20-meter track was prepared for the test. Athletes were asked to run the 20-meter distance as fast as possible. The fastest time to complete the track was recorded as a score in seconds. Microgate Witty brand photocells were placed at the start and end points to measure the time [66, 67]. The device consists of 3 parts, 2 photocell doors and tablet Photocell doors were positioned on both sides of the start and finish lines. For the test, the athlete started the photocell counter as soon as the athlete crossed the starting line. The finish photocell stopped the counter as soon as the athlete crossed the finish line.
Balance | 25 June 2023
  Y-Shaped Balance Test was used to evaluate upper extremity balance.
Right/Left Separation | 25 June 2023
  Android-based Noi Recognise App application was used for the right-left separation of the athletes. Before the test, the practice was shown to the athletes and a trial test was performed. The test was performed with a mobile device while the athletes were in a sitting position. 20 different images of hands photographed from different angles, used as standard for the test, were shown 5 seconds apart. The athlete was asked to mark which side extremity the picture he saw belonged to as quickly and accurately as possible on the screen of the application. Recognition rates and response speed obtained as a result of the test were recorded as scores on the application.
Stroop Test | 25 June 2023
  The Stroop test is widely used to evaluate cognitive functions such as selective attention and resistance to interference. There are different variations of the Stroop test. In our study, we used the Stroop Test Anchor Form, the validity and reliability of which was made by Savaş et al.
Two-Point Discrimination | 25 June 2023
  Baseline 2-point discrimination instrument was used for the two-point discrimination test. The discrimination tool was set to 5 millimeters. The tips of the instrument were touched to the most swollen area of the hypothenar region of the dominant hand, parallel to the long axis of the hand, and they were asked to say how many points they felt.
Pain Threshold Level | 25 June 2023
  Jtech Commander (JTech Medical Industries, ZEVEX Company) brand algometer device was used to evaluate the pain threshold. The most swollen point of the thenar region of the dominant hand was used to assess the pain threshold.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)